CLINICAL TRIAL: NCT06735092
Title: Investigation of the Effects of Different Types of Orthoses Used in Addition to Exercise Therapy in Lateral Elbow Tendinopathy
Brief Title: Exercise Therapy and Orthoses in Lateral Elbow Tendinopathy: Comparative Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Büşra Kültür, Master's Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-FTR-B-01
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Lateral Epicondylitis
Keywords: Exercise Therapy; Rehabilitation; Orthotic Devices; Pain; Tendinopathy
MeSH Terms: conditions — Tennis Elbow; Pain; Tendinopathy | interventions — Control Groups; Exercise

STUDY DESIGN:
Intervention Model Description: This study involves three groups with exercise therapy: one with exercise only, one with exercise in addition to an elbow orthosis, and one with exercise in addition to a wrist orthosis.
Who Masked: Participant
Masking Description: The participants in the study are blind to the group distribution and do not know the reason for their assignment to specific groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise-Only Group (Control Group) (Active Comparator): This is the control group, where the patients will only participate in an exercise program, without any additional support or devices like braces. This group helps assess the effectiveness of exercise alone compared to other interventions involving braces. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group.
  Interventions: Other: Exercise-Only Group (Control Group)
- Exercise + Forearm Counterforce Brace Group (Active Comparator): This group will focus on a combined treatment approach, including exercise therapy alongside the use of a forearm counterforce brace. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group.
  Interventions: Other: Exercise + Forearm Counterforce Brace Group
- Exercise + Wrist Brace Group (Active Comparator): This group will focus on a treatment combining exercise therapy with the use of a wrist brace. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group.
  Interventions: Other: Exercise + Wrist Brace Group

INTERVENTIONS:
Other: Exercise-Only Group (Control Group) — Participants in this group will only undergo a standardized exercise protocol. The exercises will be part of a program lasting 6 weeks, conducted 2 days per week. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group. For free-weight exercises, participants will start with weights of 0.5-1 kg, tailored to the individual. Progression will be achieved with 0.5-1 kg increments. For exercises using resistance bands, the increase in resistance will be provided by selecting the next level band color. Participants will be assessed before treatment, at the end of the 6th week, and at the end of the 12th week.
  Arms: Exercise-Only Group (Control Group)
Other: Exercise + Forearm Counterforce Brace Group — Participants in this group will undergo a standardized exercise protocol and will be provided with a counterforce forearm brace in addition to exercise therapy. The exercises will be part of a program lasting 6 weeks, conducted 2 days per week. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group. For free-weight exercises, participants will start with weights of 0.5-1 kg, tailored to the individual. Progression will be achieved with 0.5-1 kg increments. For exercises using resistance bands, the increase in resistance will be provided by selecting the next level band color. Participants will be assessed before treatment, at the end of the 6th week, and at the end of the 12th week.
  Arms: Exercise + Forearm Counterforce Brace Group
Other: Exercise + Wrist Brace Group — Participants in this group will undergo a standardized exercise protocol and will be provided with a wrist brace in addition to exercise therapy. The exercises will be part of a program lasting 6 weeks, conducted 2 days per week. A combined evidence-based exercise program consisting of wrist isometric, concentric, and eccentric exercises will be applied to the individuals in the group. For free-weight exercises, participants will start with weights of 0.5-1 kg, tailored to the individual. Progression will be achieved with 0.5-1 kg increments. For exercises using resistance bands, the increase in resistance will be provided by selecting the next level band color. Participants will be assessed before treatment, at the end of the 6th week, and at the end of the 12th week.
  Arms: Exercise + Wrist Brace Group

SUMMARY:
The aim of this study is to address the inconsistencies in the literature by investigating the effects of a forearm counterforce brace and a wrist splint, used in addition to exercise therapy, on pain, functionality, and grip strength in individuals diagnosed with lateral elbow tendinopathy, compared to those receiving exercise therapy alone.The findings aim to provide valuable insights into clinical practice by highlighting the roles of both orthosis use and exercise in the treatment of lateral elbow tendinopathy.

DETAILED DESCRIPTION:
This study will be conducted under the supervision of Istanbul University-Cerrahpasa, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation. It is designed as a randomized controlled trial and will include participants diagnosed with lateral elbow tendinopathy who meet the inclusion criteria and agree to participate. These participants will be recruited from the Orthopedics and Traumatology Clinic of Basaksehir Cam and Sakura City Hospital. Participants will be informed about the purpose, procedures, and potential risks of the study, and written informed consent forms will be obtained after the explanation. Following the signing of the informed consent forms, participants will be randomized into three groups:

1. Exercise + Counterforce Forearm Brace Group
2. Exercise + Wrist Brace Group
3. Exercise-Only Group (Control Group)

All participants will follow a standard exercise protocol. The exercises will be carried out twice a week for six weeks and will include an evidence-based combined exercise program consisting of isometric, concentric, and eccentric wrist exercises. The exercises will initially start with free weights of 0.5-1 kg, depending on the patient, with progression achieved through 0.5-1 kg weight increments. For exercises using elastic bands, resistance progression will be managed by selecting a band of higher resistance level. In addition to the exercise therapy, Group 1 participants will use a counterforce forearm brace, while Group 2 participants will use a wrist brace.

Participants will be assessed before the intervention and at the 6th and 12th weeks. A total of 45 patients diagnosed with "lateral elbow tendinopathy" by a specialist physician will be evaluated in the study. Assessments will include:

Sociodemographic characteristics and clinical status using a "Case Assessment Form" Pain levels using the "Numerical Pain Rating Scale (NPRS)" Grip strength and pain-free grip strength using a "Digital Hand Dynamometer" Functional levels using the "Patient-Rated Tennis Elbow Evaluation (PRTEE)" questionnaire developed specifically for lateral elbow tendinopathy Satisfaction with the interventions using the "Global Rating of Change Scale." The collected data will be analyzed using Statistical Package for the Social Sciences (SPSS) software.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65,
* Having a diagnosis of unilateral lateral elbow tendinopathy,
* Having at least two of the Thomsen, Maudley's, Mill's, or Cozen's tests positive during clinical examination,
* Experiencing symptoms for at least 3 months,
* Not having a systemic or chronic illness that would prevent participation in the treatment program.

Exclusion Criteria:

* A history of trauma or surgery in the relevant elbow and/or wrist,
* The presence of orthopedic and/or neurological problems in the cervical spine, shoulder joint, or wrist,
* Participation in a physiotherapy and rehabilitation program for lateral elbow tendinopathy within the last 6 months,
* Receiving any injections within the last 6 months,
* Systemic inflammation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation Questionnaire (PRTEE) | six weeks
  The Patient-Rated Tennis Elbow Evaluation (PRTEE) is a self-reported questionnaire designed to measure pain and functional limitations in individuals with lateral epicondylitis (tennis elbow). It consists of 15 items divided into two subscales: pain (5 items) and functional disability (10 items). Each item is rated on a scale from 0 (no pain or difficulty) to 10 (severe pain or difficulty), with a total score range of 0 to 100. Higher scores indicate greater pain and disability, while lower scores reflect improvement. The PRTEE is commonly used to assess treatment outcomes and track patient progress over time.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | six weeks
  The Numeric Pain Rating Scale (NPRS) is a subjective measure used to assess pain intensity. It is a 0-10 scale, where 0 indicates "no pain" and 10 represents "the worst pain imaginable." Patients are asked to rate their pain level based on this scale. A decrease in the NPRS score indicates an improvement or reduction in pain, while an increase suggests worsening pain. It is a simple and widely used tool for monitoring pain in clinical and research settings.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kültür, MSc, Principal Investigator — Istanbul University - Cerrahpasa; Derya Çelik, Prof. Dr., Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Faculty of Health Sciences, Istanbul University - Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No